CLINICAL TRIAL: NCT06084403
Title: The Efficacy of Different Volumes for Ultrasound-Guided Adductor Canal Block for Postoperative Analgesia Management After Total Knee Arthroplasty Surgery
Brief Title: Ultrasound-Guided Adductor Canal Block for Total Knee Arthroplasty Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, MD, Assoc Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCityH
Record Dates: First submitted 2023-09-30; First posted 2023-10-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Knee Disease; Knee Deformity; Knee Pain Chronic; Knee Arthropathy; Knee Osteoarthritis
Keywords: Adductor Canal Block; Total Knee Arthroplasty; Postoperative Analgesia Management
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: There are threemodels for this study. 20 ml volume adductor canal block group, 30 ml volume adductor canal block group and 40 ml volume adductor canal block group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery. Patients will be administered tenoxicam (Tilcotil 20 mg flakon) 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol (100 mg-Contramal ® ampul) will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine (Aldolan ampul 100 mg/2 ml) IV will be administered.
  Interventions: Drug: 20 ml volume adductor canal block
- 30 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery. Patients will be administered tenoxicam (Tilcotil 20 mg flakon) 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol (100 mg-Contramal ® ampul) will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine (Aldolan ampul 100 mg/2 ml) IV will be administered.
  Interventions: Drug: 30 ml volume adductor canal block
- 40 ml volume adductor canal block (Active Comparator): ACB will be performed at the end of the surgery. Patients will be administered tenoxicam (Tilcotil 20 mg flakon) 20 mg IV every 12 hours in the postoperative period. A patient controlled device prepared with 5 mg/ ml tramadol (100 mg-Contramal ® ampul) will be attached to all patients with a protocol included 10 mg bolus without infusion dose, 20 min lockout time and 4 hour limit. If the VAS score will be ≥ 4, 0,5 mg/kg-1 meperidine (Aldolan ampul 100 mg/2 ml) IV will be administered.
  Interventions: Drug: 40 ml volume adductor canal block

INTERVENTIONS:
Drug: 20 ml volume adductor canal block — ACB will be performed at the end of the surgery. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine (Buvasin %5 flakon) 20ml will be injected here.
  Arms: 20 ml volume adductor canal block
Drug: 30 ml volume adductor canal block — ACB will be performed at the end of the surgery. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine(Buvasin %5 flakon) 30ml will be injected here.
  Arms: 30 ml volume adductor canal block
Drug: 40 ml volume adductor canal block — ACB will be performed at the end of the surgery. After identifying the adductor canal, by using the in-plane technique, the probe will be placed at the mid-thigh, half the distance between the inguinal crease and the patella, for block location. The superficial femoral artery will be visualized dorsal to the sartorius muscle. Then, the probe will be removed to distally. At this level, the hyperechoic view of the saphenous nerve will be visualized lateral and anterior to the artery in the subsartorial region. 5 mL of saline will be injected to confirm the proper injection site, and then a dose of 0.25% bupivacaine(Buvasin %5 flakon) 40ml will be injected here.
  Arms: 40 ml volume adductor canal block

SUMMARY:
The ultrasound-guided selective blockade of the saphenous nerve in the adductor canal provides effective analgesia and reduces postoperative pain in patients undergoing arthroscopic medial meniscectomy. Selective blockade of the saphenous nerve in the adductor canal provides effective analgesia without quadriceps muscle weakness. It has been shown that the adductor canal block (ACB) block increases the spread of local anesthetics in a distal and proximal way. Therefore, the proximal spread of local anesthetics may cause possible quadriceps weakness. The distal spread of local anesthetics may increase analgesic effect via sciatic nerve. The different volumes for ACB is a topic of discussion. The aim of this study is to compare the different volumes of US-guided ACB performing for postoperative analgesia management after total knee arthroplasty surgery.

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most common orthopedic procedures. Patients may complain severe pain due to the surgical trauma and the prosthesis. Opioid agents are commonly used for analgesia management. However, opioids have adverse effects such as nausea, vomiting, sedation and respiratory depression. Peripheral nerve blocks such as femoral block, adductor canal block (ACB) may be performed to reduce opioid consumption and opioid-related side effects.

Selective blockade of the saphenous nerve in the adductor canal for knee surgery provides effective analgesia without quadriceps muscle weakness. This is an important advantage of ACB since it there is no motor blockade in the postoperative period. Blocking of the motor branches leads to delaying of the mobilization and it increases the patient's falling risk. ACB, targets the saphenous nerve and the vastus medialis branch which are the two largest sensorial nerves of the femoral nerve that innervates the knee. ACB blocks the articular branches of the obturator nerve at the same time. Since the ACB is performed at the distal site of thigh it does not target majority of the efferent branches of the quadriceps muscle, therefore the strength of this muscle may not be affected. ACB is usually performed with a volume of 10-30 ml and studies may be needed including different volumes to understand its effectiveness.

The aim of this study is to compare the different volumes (20 ml, 30 ml, and 40 ml) of US-guided ACB for postoperative analgesia management after total knee arthroplasty. The primary aim is to compare postoperative opioid consumption and the secondary aim is to evaluate postoperative pain scores (VAS), motor blockage, the first mobilization time, and adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II-III
* Scheduled for total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* history of bleeding diathesis
* receiving anticoagulant treatment,
* known local anesthetics and opioid allergy,
* infection of the skin at the site of the needle puncture,
* pregnancy or lactation,
* patients who do not accept the procedur

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Opioid consumption will be recorded at the first 48 hours period postoperatively
  The primary aim is to compare perioperative and postoperative opioid consumption.
  Opioid consumption will be recorded at the first 48 hours period postoperatively.
  (postoperative 0-8, 8-16, 16-24, 24-48 hours)

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Patients will be evaluated at the first 48 hours period postoperatively
  Postoperative 48 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16, 24 and 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Mürsel Ekinci, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not share IPD

REFERENCES:
- [Background] Guven Kose S, Kose HC, Arslan G, Eler Cevik B, Tulgar S. Evaluation of ultrasound-guided adductor canal block with two different concentration of bupivacaine in arthroscopic knee surgery: A feasibility study. Int J Clin Pract. 2021 Nov;75(11):e14747. doi: 10.1111/ijcp.14747. Epub 2021 Sep 3. PMID 34428334
- [Background] Ekinci M, Ciftci B, Demiraran Y, Celik EC, Yayik M, Omur B, Kuyucu E, Atalay YO. A comparison of adductor canal block before and after thigh tourniquet during knee arthroscopy: a randomized, blinded study. Korean J Anesthesiol. 2021 Dec;74(6):514-521. doi: 10.4097/kja.21040. Epub 2021 May 13. PMID 33984219
- [Background] Frassanito L, Vergari A, Nestorini R, Cerulli G, Placella G, Pace V, Rossi M. Enhanced recovery after surgery (ERAS) in hip and knee replacement surgery: description of a multidisciplinary program to improve management of the patients undergoing major orthopedic surgery. Musculoskelet Surg. 2020 Apr;104(1):87-92. doi: 10.1007/s12306-019-00603-4. Epub 2019 May 3. PMID 31054080
- [Derived] Ekinci M, Kaciroglu A, Dikici M, Yildiz Eglen M, Bayrak F, Aydogmus I, Celik EC, Ciftci B. Effects of ultrasound-guided adductor canal block at different volumes on postoperative analgesia management in patients undergoing total knee arthroplasty: a prospective clinical study. BMC Anesthesiol. 2025 Oct 20;25(1):510. doi: 10.1186/s12871-025-03383-6. PMID 41116173